CLINICAL TRIAL: NCT05196113
Title: sipIT2: Improving Adherence to Fluid Intake Guidelines for Kidney Stone Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, David Conroy, Bickner Chair of Kinesiology and Professor of Kinesiology, School of Kinesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00015540; R01DK124469 (NIH)
Record Dates: First submitted 2021-12-03; First posted 2022-01-19 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sipIT (Experimental): Participants receive education and a digital tool to monitor their fluid intake and remind them when they have lapsed in regular fluid intake.
  Interventions: Behavioral: sipIT
- Control (No Intervention): Participants receive usual care (i.e., education about fluid intake guidelines and encouragement to meet those guidelines).

INTERVENTIONS:
Behavioral: sipIT — Participants receive education and digital tools to monitor their fluid intake and just-in-time text messages to remind them when they have lapsed in regular fluid intake.
  Arms: sipIT

SUMMARY:
The purpose of this study is to examine the feasibility of using sipIT tools (i.e., wrist-worn sensors, smart water bottles, mobile applications) to increase compliance with physician-recommended fluid consumption guidelines in participants with a history of urolithiasis.

DETAILED DESCRIPTION:
The study uses a randomized controlled trial design with a 12-month intervention period and outcome assessments at baseline, 1, 3, and 12 months. Participants will be randomly assigned to groups. Both groups will receive usual care which involves education about fluid intake guidelines and encouragement to adhere to those guidelines from a clinician. The intervention group will additionally receive the sipIT intervention comprising a semi-automated fluid intake tracking system and context-sensitive, just-in-time notifications reminding them to drink.

ELIGIBILITY:
Inclusion Criteria:

* previous diagnosis of symptomatic kidney stone in past 5 yrs
* 24-hr urine volume ≤ 2.0 L/day,
* age 18 or older,
* own iOS or Android smartphone,
* proficient in English language,
* capable of providing informed consent, and
* willing to use a Fitbit smartwatch, connected water bottle, and mobile app for the study every day for a year, and receive text messages reminder to drink.

Exclusion Criteria:

* previous diagnosis with cystine stone,
* pregnant or planning to become pregnant in the next 12 months,
* concurrently participating in another study involving fluid intake or diet,
* plan to have surgery or relocate outside the area within the next year
* co-morbidities that preclude high fluid intake, conditions with high fluid losses (e.g., congestive heart failure, bariatric surgery, GI tract ostomy, short gut syndrome, chronic diarrhea including patients with ulcerative colitis/Crohn's disease, hyponatremia), or conditions that preclude ability to collect 24-hour urine (severe urinary incontinence),
* active medical treatments that would impair protocol compliance,
* chronic use of lithium, or
* psychiatric conditions impairing compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
24-hr urine volume | 12 months
  Change in urine volume from baseline

SECONDARY OUTCOMES:
24-hr urine volume | 1 month and 3 months
  Change in urine volume from baseline
Urine supersaturations | 1 month, 3 months, and 12 months
  Change in supersaturations of common stone-forming salts from baseline to 1/3/12 months
Habit strength for fluid intake | 3 months, and 12 months
  Change in habit by the 4-item Self-Report Behavioural Automaticity Index (Gardner, Abraham, Lally & de Bruijn, 2012, Int J Beh Nutr Phys Act; baseline to 3/12 months). Responses will be averaged so scores range from 1 (strongly disagree) to 7 (strongly agree) with higher scores indicating stronger habits for fluid intake.
Past-week fluid intake | 3 months, and 12 months
  Change in past-week volume of fluid intake from baseline to 3/12 months

CONTACTS AND LOCATIONS:
Overall Officials: David E Conroy, PhD, Principal Investigator — University of Michigan; Necole M Streeper, MD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Penn State Hershey Medical Center, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conroy DE, Marks J, Cutshaw A, Ram N, Thomaz E, Streeper NM. Promoting fluid intake to increase urine volume for kidney stone prevention: Protocol for a randomized controlled efficacy trial of the sipIT intervention. Contemp Clin Trials. 2024 Mar;138:107454. doi: 10.1016/j.cct.2024.107454. Epub 2024 Jan 20. PMID 38253254

DOCUMENTS (1):
  • Informed Consent Form (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT05196113/ICF_000.pdf